CLINICAL TRIAL: NCT00143065
Title: Feasibility/Phase II Trial of Fludarabine, Rituximab, and Alemtuzumab for Previously Treated B-Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL)
Brief Title: Fludarabine, Rituximab, and Alemtuzumab for B-Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, John Byrd, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0404
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Lymphoma, Small Lymphocytic; Lymphocytic Leukemia, Chronic
Keywords: Antigens, CD5; Antigens, CD19; Antigens, CD20
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine; fludarabine phosphate; Rituximab; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fludarabine — 25 mg/m2/day for 5 days every 28 days (Week 2,6,10,14, 18,and 22) will be administered by IV over 10-30 minutes. (Fludarabine should be given AFTER rituximab on all days on which both drugs will be administered.)
  Other Names: Fludara
Drug: Rituximab — Day 1, week 2 of cycle 1 rituximab 100 mg will be administered by IV, without dose escalation, over 4 hours (rate: 25 mg/hr). Day 3, week 2 of cycle 1 rituximab 375 mg/m2 will be administered by IV. Rituximab can be administered at 50 mg/hr. If hypersensitivity or infusion related events do not occur, the infusion rate will be escalated in 50 mg/hr increments every 30 minutes to a maximum of 400 mg/hr.
  * On Day 5, week 2 of cycle 1 rituximab 375 mg/m2 will be administered by IV. Rituximab can be administered at 100 mg/hr. If hypersensitivity or infusion related events do not occur, the infusion rate will be escalated in 100 mg/hr increments every 30 minutes to a maximum of 400 mg/hr.
  * Rituximab 375 mg/m2 will be repeated on Day 1 of Week 6, 10, 14, 18, and 22. During these treatments, acetaminophen and diphenhydramine prophylactic treatment is left to the discretion of the treating physician.
  Other Names: Rituxan
Drug: Alemtuzumab — The dose of alemtuzumab will be escalated during Week 1 of therapy. On Day 1 of Week 1, a dose of 3 mg should be administered IV over 2-hours. If this dose is well tolerated(grade 2 or less infusion or skin related toxicity), then the dose on Day 2 can be increased to 10 mg IV over 2 hours. If this dose is well tolerated, then the dose on Day 3 will be increased to 30 mg IV over 2-hours, and if tolerated, then day 5 and all subsequent alemtuzumab doses will be 30 mg. Vital signs (blood pressure, pulse, respiration rate,temperature, and O2 saturation) and skin assessment should be assessed at baseline, 1-hour, and 1-hour post administration during week 1 and 2. Following successful escalation to 30 mg of alemtuzumab, all subsequent doses of alemtuzumab will be 30 mg administered on the second day of fludarabine therapy (week 2,6,10,14,18,and 22).
  Other Names: Campath

SUMMARY:
This purpose of this study is to assess the toxicity and the rate of complete and overall response using fludarabine, rituximab, and alemtuzumab to treat patients with B-chronic lymphocytic leukemia or small lymphocytic leukemia who have received previous treatment.

DETAILED DESCRIPTION:
Immunotherapy, or treatments that work by boosting immune function in the body, such as monoclonal antibodies have shown some efficacy against different types of leukemia. Researchers have learned to manufacture antibodies outside of the human body that can bind to specific targets in cancer cells. Monoclonal antibodies are designed to recognize different proteins on specific cancer cells. The current study combines two monoclonal antibodies, rituximab and fludarabine. Rituximab attaches to a protein called the CD20 antigen that is found almost exclusively on the surface of B-cells with leukemia. Once rituximab attaches to the protein, the immune system activates to kill the malignant B-cells. Alemtuzumab works in a similar way by attaching with the CD25 antigen and also has activity in patients with p53 gene mutations. Previous studies indicate that both rituximab and alemtuzumab separately have some efficacy against lymphocytic leukemia. Research has also shown that fludarabine works against the disease. Rituximab and fludarabine in combination appear to have a high response rate in patients. Researchers are seeking to improve efficacy data by adding alemtuzumab to the combination of rituximab and fludarabine in this study.

This study will evaluate the safety and efficacy of fludarabine, rituximab, and alemtuzumab in patients with previously treated B-cell lymphocytic leukemia and small lymphocytic leukemia. Blood and bone marrow tests will assess genetic features associated with response to therapy, immune recovery, mechanisms of alemtuzumab's signaling, routes of drug resistance, and traces of residual disease following complete response in patients.

Patients in this study will receive fludarabine, rituximab, and alemtuzumab. These drugs will be administered through intravenous infusions. The treatment period will last 22 weeks. Fludarabine will not be given during week one, 5 days during week 2, and 5 days during weeks 6, 10, 14, 18, and 22. Rituximab will not be given during week one, 3 times the second week, and day one of weeks 6, 10, 14, 18, and 22. Alemtuzumab will be given 3 times during week one, once during week 2, and day 2 of weeks 6, 10, 14, 18, and 22. The dosage amount of rituximab and alemtuzumab will be increased depending upon the degree of side effects. Several tests and exams will be given throughout the study to closely monitor patients. Treatments will be discontinued due to disease growth or unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Must have B-CLL/SLL
* active disease
* >=1 prior systemic therapy
* ECOG PS 0-2.

Exclusion Criteria:

* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-08; Primary Completion 2007-02 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Assess the rate of complete (CR) and overall response (ORR) using fludarabine, rituximab, and alemtuzumab | 2005-present

SECONDARY OUTCOMES:
Assess toxicity of this regimen. | 2005-present

CONTACTS AND LOCATIONS:
Overall Officials: John C. Byrd, M.D., Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu/.